CLINICAL TRIAL: NCT01791218
Title: Concomitant Pulmonary Vein Isolation in Treatment of Paroxysmal Atrial Fibrillation Patients Undergoing Elective Coronary Artery Bypass Grafting and Aortic Valve Replacement for Aortic Stenosis: a Prospective Study
Brief Title: Surgical Pulmonary Vein Isolation Efficiency Study
Acronym: FIN-PVI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Not enough patients for study arms
Sponsor: Kuopio University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KUH5101071
Record Dates: First submitted 2013-02-12; First posted 2013-02-13 (Estimated); Last update posted 2020-09-02 (Actual); Status verified 2020-09

CONDITIONS: Paroxysmal Atrial Fibrillation; Coronary Artery Disease
Keywords: Pulmonary vein isolation; Paroxysmal atrial fibrillation; Quality of life
MeSH Terms: conditions — Atrial Fibrillation; Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CABG, AVR or CABG+AVR and PVI (Experimental): Coronary artery bypass (CABG), aortic valve replacement for aortic stenosis (AVR) or combination (CABG+AVR) using cardio-pulmonary bypass (CBP) and occlusion. Concomitant pulmonary vein isolation (PVI) in CBP prior to occlusion and CABG
  Interventions: Procedure: CABG, AVR or CABG+AVR and PVI
- CABG, AVR or CABG+AVR (Active Comparator): Coronary artery bypass (CABG), aortic valve replacement for aortic stenosis(AVR) or combination(CABG+AVR) using cardio-pulmonary bypass (CBP) and occlusion. No operative procedures for the treatment of atrial fibrillation
  Interventions: Procedure: CABG, AVR or CABG+AVR

INTERVENTIONS:
Procedure: CABG, AVR or CABG+AVR and PVI
  Arms: CABG, AVR or CABG+AVR and PVI
Procedure: CABG, AVR or CABG+AVR
  Arms: CABG, AVR or CABG+AVR

SUMMARY:
A substantial proportion of patients undergoing elective coronary artery bypass grafting have a history of paroxysmal atrial fibrillation. Paroxysmal atrial fibrillation has adverse short-and long term postoperative effects. Pulmonary vein isolation (PVI) seems to be effective treatment for paroxysmal atrial fibrillation. PVI can be done concomitantly with coronary artery bypass grafting, aortic valve replacement for aortic stenosis and combination of them. Procedure is well defined and safe.

There is a lack of convincing evidence of the effect on postoperative atrial fibrillation burden, quality of life and symptoms especially in correlation with atrial fibrillation paroxysms.

ELIGIBILITY:
Inclusion Criteria:

* American College of Cardiology (ACC)/ American Heart Association (AHA) -Indications for CABG
* At least 2 ECG-verified (12-channel ECG, Holter telemetry) symptomatic paroxysmal atrial fibrillation episodes within last 12 months
* Duration of the atrial fibrillation episode must not exceed 1 week and it must reverse to sinus rhythm spontaneously or by cardioversion
* written and verbal consent

Exclusion Criteria:

* Prior cardiac surgery
* Active pacemaker treatment
* Active anti-arrhythmic treatment(AAD) class I and III
* Contraindication to oral anticoagulant/heparin treatment
* Ejection fraction less than 30 % (EF < 30 %)assessed by transthoracic echocardiography
* Left atrial diameter less than 55mm assessed by transthoracic echocardiography
* Renal insufficiency requiring dialysis
* Heart valve disease requiring invasive treatment
* Heart anomaly requiring regular controls and/or invasive treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2012-11; Primary Completion 2020-09 (Actual); Study Completion 2020-09 (Actual)

PRIMARY OUTCOMES:
Atrial fibrillation burden | Within one year after operative treatment
  Atrial fibrillation burden is defined as the amount of atrial fibrillation on one week Holter monitoring
Freedom of symptomatic and asymptomatic atrial fibrillation after surgery | Within one year after operative treatment
  Atrial fibrillation is defined as atrial fibrillation paroxysm lasting at least 60 seconds.
  Freedom of atrial fibrillation is defined as duration of atrial fibrillation less than 0,5% of the one week Holter monitoring

SECONDARY OUTCOMES:
Compare quality of life (QOL) and symptoms, correlation of symptoms with atrial fibrillation | Within one year after operative treatment
Adverse events after surgery in both arms | Within one year after operative treatment
Anti-arrhythmic treatment after surgery | Within one year after treatment
Hospitalization due to atrial fibrillation after surgery | Within one year after operative treatment
Cardioversion for the treatment of atrial fibrillation after surgery | Within one year after operative treatment
Other cardiovascular related events: death, stroke, cardiac infarction, need for revascularization and bleeding | Within one year after operative treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Kuopio University Hospital, Kuopio, Eastern Finland, Finland